CLINICAL TRIAL: NCT03621137
Title: TREAT NL (TREatment of ATopic Eczema, the Netherlands) Registry
Brief Title: TREAT NL (TREatment of ATopic Eczema, the Netherlands) Registry: Dutch National Registry for Patients With Moderate-to-severe Atopic Eczema on Photo- or Systemic Therapies
Acronym: TREAT NL
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Angela Bosma, Co-investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: TREAT NL registry
Record Dates: First submitted 2018-07-06; First posted 2018-08-08 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Moderate-to-severe Atopic Eczema
Keywords: Atopic Eczema; Atopic Dermatitis; Registries; Systemic therapies; Off-label use; Phototherapy; Child; Adult
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — TREAT NL biobank substudy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with moderate-to-severe atopic eczema: Adult and pediatric patients that start treatment with phototherapy or systemic immunomodulating therapy for their atopic eczema
  Interventions: Other: No study-specific intervention

INTERVENTIONS:
Other: No study-specific intervention — Treatment of atopic eczema with phototherapy or systemic immunomodulating therapy according to usual clinical practice

SUMMARY:
The TREAT NL (TREatment of ATopic eczema, the Netherlands) registry is a national registry for children and adults with moderate-to-severe atopic eczema aiming to gather data on their prescribed photo- and systemic immunomodulating therapies. Atopic eczema is a common, chronic, itchy, inflammatory skin disease that can have a major impact on the quality of life of patients and their immediate surroundings.

Serious atopic eczema patients are treated by means of photo- or systemic immunomodulating therapy. Of these mostly off-label applied therapies, there is insufficient evidence on the short and long term for their effectiveness, safety and cost-effectiveness. Moreover, good comparative research and real-life data are lacking. With the arrival of new expensive treatments it is crucial to get insight into these treatments in order to improve quality of care.

By means of a prospective registry these data can be collected and help to obtain information for clinical practice, for answering research questions, for reducing costs and implementing the results by guidelines and decision aids.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of atopic eczema, based on the U.K. working party's diagnostic criteria;
* Starts with any type of phototherapy (e.g. UVB) or systemic immunomodulating therapy (e.g. cyclosporin, systemic glucocorticosteroids, azathioprine, methotrexate, mycophenolic acid, dupilumab);
* Has voluntarily signed and dated an informed consent prior to any study related procedure or has a legal representative to do so and is willing to comply with the requirements of this study protocol.

Exclusion Criteria:

* Patient uses only (systemic) antibiotics or antihistamines;
* Patient starts with systemic immunomodulating therapy for another indication than atopic eczema;
* Insufficient understanding of the study by the patient or parent/legal representative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of participating centres that meet the predefined in- and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in EASI (Eczema Area and Severity Index) score | 5 years
  Investigator-assessed outcome measure for disease severity at physical examination
Mean change in IGA (Investigator's Global Assessment) score | 5 years
  Investigator-assessed outcome measure for global disease severity
Mean change in POEM (Patient-Oriented Eczema Measure) score | 5 years
  Patient-reported outcome measure for symptoms of atopic eczema
Mean change in PGA (Patient's Global Assessment) score | 5 years
  Patient-reported outcome measure for global disease severity
Mean change in DLQI (Dermatology Life Quality Index) score | 5 years
  Patient-reported outcome measure for skin-related quality of life
Mean time to reach a change in EASI (Eczema Area and Severity Index) score of 50% | 5 years
  Investigator-assessed outcome measure for disease severity at physical examination
The occurrence of severe adverse events | 5 years
  Any undesirable experience of severe nature occurring to a subject is reported
Drug survival of the therapies | 5 years
  Assessment of the duration until discontinuation of a drug together with the reason thereof

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis I. Spuls, prof.dr., Principal Investigator — Department of Dermatology, Amsterdam University Medical Centres, University of Amsterdam, Research Institute Amsterdam Public Health and Amsterdam Infection and Immunity Institute, Amsterdam, The Netherlands
Locations (1):
- Department of Dermatology, Amsterdam University Medical Centres, University of Amsterdam, Research Institute Amsterdam Public Health and Amsterdam Infection and Immunity Institute, Amsterdam, The Netherlands, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gerbens LA, Boyce AE, Wall D, Barbarot S, de Booij RJ, Deleuran M, Middelkamp-Hup MA, Roberts A, Vestergaard C, Weidinger S, Apfelbacher CJ, Irvine AD, Schmitt J, Williamson PR, Spuls PI, Flohr C. TREatment of ATopic eczema (TREAT) Registry Taskforce: protocol for an international Delphi exercise to identify a core set of domains and domain items for national atopic eczema registries. Trials. 2017 Feb 27;18(1):87. doi: 10.1186/s13063-016-1765-7. PMID 28241851
- [Background] Spuls PI, Gerbens LAA, Apfelbacher CJ, Wall D, Arents BWM, Barbarot S, Roberts A, Deleuran M, Middelkamp-Hup MA, Vestergaard C, Weidinger S, Schmitt J, Irvine AD, Flohr C. The International TREatment of ATopic Eczema (TREAT) Registry Taskforce: An Initiative to Harmonize Data Collection across National Atopic Eczema Photo- and Systemic Therapy Registries. J Invest Dermatol. 2017 Sep;137(9):2014-2016. doi: 10.1016/j.jid.2017.05.014. Epub 2017 May 27. No abstract available. PMID 28558913
- [Background] Gerbens LAA, Apfelbacher CJ, Irvine AD, Barbarot S, de Booij RJ, Boyce AE, Deleuran M, Eichenfield LF, Hof MH, Middelkamp-Hup MA, Roberts A, Schmitt J, Vestergaard C, Wall D, Weidinger S, Williamson PR, Flohr C, Spuls PI; international TREAT Registry Taskforce. TREatment of ATopic eczema (TREAT) Registry Taskforce: an international Delphi exercise to identify a core set of domains and domain items for national atopic eczema photo- and systemic therapy registries. Br J Dermatol. 2019 Apr;180(4):790-801. doi: 10.1111/bjd.16714. Epub 2018 Aug 3. PMID 29761486
- See also: Website of the international TREAT Registry Taskforce — https://treat-registry-taskforce.org/